CLINICAL TRIAL: NCT05881811
Title: An Open-label Phase I Study to Evaluate the Drug-drug Interaction of HSK16149 Capsule With Probenecid Tablets or Cimetidine Tablets in Healthy Subjects
Brief Title: The Drug-drug Interaction of HSK16149 Capsule With Probenecid Tablets or Cimetidine Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HSK16149-105
Record Dates: First submitted 2023-05-16; First posted 2023-05-31 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: PHN - Post-Herpetic Neuritis
MeSH Terms: interventions — Cimetidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 (Experimental): Period 1: HSK16149 single dose on D1, 40mg, fasted; Period 2: HSK16149 single dose on D2, 40mg, fasted; Probenecid QID (500mg) on D1~D4. HSK16149 would be administered 2 hours after the first dose of probenecid on D2.
  Interventions: Drug: HSK16149，probenecid, cimetidine
- A2 (Experimental): Period 1: HSK16149 single dose on D2, 40mg, fasted；probenecid QID (500mg) on D1~D4. HSK16149 would be administered 2 hours after the first dose of Probenecid on D2.
  Period 2: HSK16149 single dose on D1, 40mg, fasted;
  Interventions: Drug: HSK16149，probenecid, cimetidine
- B1 (Experimental): Period 1: HSK16149 single dose on D1, 40mg, fasted; Period 2: HSK16149 single dose on D2, 40mg, fasted; Cimetidine QID (200mg) on D1~D4. HSK16149 would be administered 1 hour after the first dose of Cimetidine on D2.
  Interventions: Drug: HSK16149，probenecid, cimetidine
- B2 (Experimental): Period 1: HSK16149 single dose on D2, 40mg, fasted; Cimetidine QID (200mg) on D1~D4. HSK16149 would be administered 1 hour after the first dose of Cimetidine on D2.
  Period 2: HSK16149 single dose on D1, 40mg, fasted;
  Interventions: Drug: HSK16149，probenecid, cimetidine

INTERVENTIONS:
Drug: HSK16149，probenecid, cimetidine — 40mg HSK16149 single dose, fasted; 500mg probenecid QID from D1~D4 200mg cimetidine QID from D1~D4

SUMMARY:
This study is a single-center, open-label, crossover study, conducted in healthy Chinese populations, and plans to enroll 48 healthy adult subjects (male and female).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
2. 18 years to 50 years (inclusive), male and female;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-28 kg/m2 (inclusive);
4. Physical examination, vital sign measurements results were deemed appropriate by the investigator;
5. Not in use of any drug within 2 weeks prior to screening;

7. Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration.

Exclusion Criteria:

1. Have an allergic history to the main ingredients and/or any auxiliary materials in the research preparation, allergic diseases or allergies, or allergic history to pregabalin or gabapentin, or allergic history to pregabalin or gabapentin or sulfonamides;
2. Have special requirements for diet and cannot follow the unified diet;
3. The abnormal results of 12-lead electrocardiogram (ECG), chest X-ray (positive position) and routine laboratory tests (blood routine, blood biochemistry, urine routine and coagulation function) during the screening period have clinical significance and are judged by the researchers to be unsuitable to participate in this experiment;
4. In the screening period, male QTcF>450 milliseconds (msec) and female QTcF>470 milliseconds (msec);
5. dizziness or vertigo with clinical significance and requiring medical intervention, or history of inner ear diseases known to cause dizziness or vertigo;
6. Insomnia, anxiety disorder, depression disorder or other mental disorders requiring medical intervention;
7. Use any caffeinated food or drink (coffee, tea, cola, chocolate, etc.) within 48 hours before the first administration of the experimental drug, or disagree with the prohibition of using any caffeinated food or drink during the trial；
8. Suffering from or having suffered from major diseases of cardiovascular system, respiratory system, digestive system, urinary system, hematology, endocrine system, immunity system, skin system or nervous system, including acute diseases or major surgical operations within 3 months before screening；
9. Suffering from or having suffered from diseases of gastrointestinal tract, liver, kidney or other known diseases that interfere with drug absorption, distribution, metabolism or excretion;
10. Blood donation or blood loss of ≥400 mL or more within 3 months before the first administration of the experimental drug;
11. Any drugs that inhibit or induce liver drug metabolizing enzymes have been used within 28 days before the first administration of experimental drugs (such as barbiturates, carbamazepine, phenytoin, glucocorticoid and omeprazole; Inhibitor serotonin reuptake inhibitor (SSRI) antidepressants, cimetidine, diltiazem macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines), or any prescription drugs, over-the-counter drugs, Chinese patent medicines and herbs other than the above drugs were taken orally within 14 days before the administration of the experimental drugs;
12. have participated in clinical trials of other drugs within 3 months before the first administration of experimental drugs;
13. Use any live vaccine within 28 days before the first administration of experimental drugs;
14. At present, they are or have been drug users, or they are positive in drug abuse screening (screening items include: morphine, tetrahydrocannabinol, methamphetamine, methylenedioxyamphetamine, ketamine and cocaine);
15. Regular drinkers within 3 months before the first administration of the experimental drug, that is, those who drink more than 14 units of alcohol per week (1 unit =10g pure alcohol, or 285mL beer [4.9% Alc./Vol] or 30 mL spirits [40% Alc./Vol] or 100 mL wine [12% Alc./Vol]), or the alcohol breath test is positive；
16. Smoking more than 5 cigarettes per day (or using a considerable amount of nicotine-containing products) within 3 months before the first administration of experimental drugs, or failing to comply with the smoking ban during the trial;
17. One or more of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, syphilis antibody or human immunodeficiency virus (HIV) antibody are positive during the screening period;
18. Have any history of malignant tumor in recent 10 years;
19. pregnant or lactating women;
20. The estimated glomerular filtration rate (eGFR) during the screening period is clinically significant or has a history of kidney calculi's disease and kidney disease;
21. Subjects with poor compliance or other factors that are not suitable for participating in this experiment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Cmax | From the start to 72 hours after administration
  The maximun plasma concentration of HSK16149
AUC0-t | From the start to 72 hours after administration
  Area under the concentration-time curve from time zero to time of last quantifiable concentration
AUC0-inf | From the start to 72 hours after administration
  Area under the concentration-time curve from time zero extrapolated to infinite time

SECONDARY OUTCOMES:
Tmax | From the start to 72 hours after administration
  Time of maximum concentration
t1/2 | From the start to 72 hours after administration
  half life
Vz | From the start to 72 hours after administration
  Volume of distribution associated with the terminal phase
CL | From the start to 72 hours after administration
  Plasma clearance
Ae | From the start to 72 hours after administration
  Cumulative urinary recovery of unchanged drug
Fe | From the start to 72 hours after administration
  Cumulative urinary recovery fraction of unchanged drug
CLr | From the start to 72 hours after administration
  Renal clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hoispital, Beijing, China